CLINICAL TRIAL: NCT03507959
Title: Components of Placebo Effects in Sadness (COPES): An Experimental Study Comparing Deceptive and Non-deceptive Placebos
Brief Title: Components of Placebo Effects in Sadness
Acronym: COPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-40v
Record Dates: First submitted 2018-03-07; First posted 2018-04-25 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Dysphoric Mood

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of five experimental groups in parallel for the duration of the study
Who Masked: Investigator
Masking Description: With regard to the four treatment groups, the investigator is not aware which experimental condition participants were allocated to. Regarding the control group, masking is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- OLP scientifically-objective (Experimental): Participants are informed that they are about to take a placebo. The rationale for the effectivity of placebos is explained in a scientifically-objective manner.
  Interventions: Other: OLP scientifically-objective
- OLP personally-affective (Experimental): Participants are informed that they are about to take a placebo. The rationale for the effectivity of placebos is explained in a personally-affective manner.
  Interventions: Other: OLP personally-affective
- DP scientifically-objective (Experimental): Participants are informed that they are about to take an effective antidepressant. The rationale for the effectivity of the antidepressant is explained in a scientifically-objective manner.
  Interventions: Other: DP scientifically-objective
- DP personally-affective (Experimental): Participants are informed that they are about to take an effective antidepressant. The rationale for the effectivity of the antidepressant is explained in a personally-affective manner.
  Interventions: Other: DP personally-affective
- Control group (No Intervention): This group does not take the nasal spray.

INTERVENTIONS:
Other: OLP scientifically-objective — Participants are informed that they are about to take a placebo. The rationale for the effectivity of placebos is explained in a scientifically-objective manner.
  Arms: OLP scientifically-objective
Other: OLP personally-affective — Participants are informed that they are about to take a placebo. The rationale for the effectivity of placebos is explained in a personally-affective manner.
  Arms: OLP personally-affective
Other: DP scientifically-objective — Participants are informed that they are about to take an effective antidepressant. The rationale for the effectivity of the antidepressant is explained in a scientifically-objective manner.
  Arms: DP scientifically-objective
Other: DP personally-affective — Participants are informed that they are about to take an effective antidepressant. The rationale for the effectivity of the antidepressant is explained in a personally-affective manner.
  Arms: DP personally-affective

SUMMARY:
Research has shown that placebo effects contribute substantially to clinical outcomes. Recent evidence suggests that placebos remain effective even if they are openly described as placebos (so-called Open-Label Placebos). In this study, the investigators examine components of open-label placebos and traditional deceptive placebos in an experimental study investigating sadness.

DETAILED DESCRIPTION:
A growing body of research has indicated that placebos contribute substantially to clinical outcomes. Yet, the implementation of deceptive placebos in clinical practice is incompatible with key principles of openness and patient autonomy. However, recent research suggests that placebos remain effective even if they openly described as placebos (so-called Open-Label Placebos (OLP)), hence questioning the necessity of deception in clinical trials.

However, comparisons between OLP and deceptive placebos (DP) with regard to their particular mechanisms are lacking. Therefore, the current study aims to identify components of OLP and DP. For this purpose, experimentally induced sadness is examined using a standardized paradigm which has previously been developed by our working group. In particular, healthy volunteers are informed that a new application method for a well-known antidepressant would be tested. Sadness is assessed before and after receiving a nasal spray. Two experimental groups (DP groups) are informed that they would receive an antidepressant nasal spray, another two experimental groups (OLP groups) are informed that they would receive a placebo. In fact, all nasal sprays are active placebos inducing prickling nasal sensations (sesame oil with 0.014% capsaicin). In addition to the factor "Transparency" (DP vs. OLP), the instruction is experimentally varied, with which the substance is administered (scientifically-objective vs. personally-affective), resulting in a 2x2 design. Further, there is an additional fifth group receiving no intervention. The primary outcome is self-rated sadness after taking the nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years
* no mental disorder or physical disease
* sufficient German language knowledge

Exclusion Criteria:

* intake of psychopharmacological drugs
* intake of illegal drugs in the last two weeks
* consumption of alcohol in the last twelve hours
* allergy to capsaicin or sesame

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS) | Baseline and 45 minutes
  Change of self-rated sadness

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kube, PhD, Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps-University of Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared